CLINICAL TRIAL: NCT03239717
Title: The Metabolic Response to Reduced Branched-chain Amino Acids in Humans
Acronym: SOAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017-0099; Protocol Version 2/23/2021 (Other: UW Madison); A534245 (Other: UW Madison); SMPH\MEDICINE\ENDOCRINOL (Other: UW Madison)
Record Dates: First submitted 2017-05-16; First posted 2017-08-04 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Obesity; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein powder (Placebo Comparator): Participants in the Placebo Arm will replace two-thirds of participants dietary protein intake with meal replacement beverages utilizing a complete protein powder.
  Interventions: Other: Whey protein powder
- Experimental (Experimental): Participants in the Experimental Arm will replace two-thirds of participants dietary protein intake with BCAD2 (Mead Johnson), a BCAA-free medical food.
  Interventions: Other: BCAD2

INTERVENTIONS:
Other: Whey protein powder — Participants in the Control Arm will replace two-thirds of participants dietary protein intake with a commercially available whey protein powder.
  Arms: Whey protein powder
Other: BCAD2 — Participants in the Experimental Arm will replace two-thirds of participants dietary protein intake with BCAD2 (Mead Johnson), a BCAA-free medical food.
  Arms: Experimental

SUMMARY:
Branched-chain amino acids (BCAAs) are essential nutrients that the body obtains from proteins found in food, especially meat, diary products, and legumes. Data from rodent studies suggest that reduction of dietary BCAAs will promote fat mass loss and improved control of blood glucose. The purpose of this study is to test if reduction of dietary BCAAs without reducing calorie intake will lead to similar metabolic benefits in humans. Here the investigators test the feasibility of reducing dietary BCAAs using BCAA-free meal replacement beverages for two months.

DETAILED DESCRIPTION:
This study, which will be completed over three months, involves replacing two meals a day with meal replacement beverages for two months, with a one month follow-up visit. These beverages will be made up by subjects using either a complete protein powder or BCAD2, a BCAA-free medical food. Participants will complete food diaries at baseline and at one month intervals during the study, and compliance will be assessed via food diaries, weekly telephone contact, and measuring returned food powder.

ELIGIBILITY:
Inclusion Criteria:

1. Male between the age of 35 - 65
2. BMI between 28 - 35 (mildly obese/overweight)
3. Fasting glucose level of 101 - 125 mg/dL
4. Able and willing to give written informed consent
5. Stable weight (within 5 lbs. for at least 3 months)
6. Not taking (or willing to cease taking) over the counter vitamin/mineral supplements
7. Not planning to begin an exercise or diet program

Exclusion Criteria:

1. Female
2. Outside required age range of 35 - 65
3. BMI not within range of 28 - 35
4. Fasting glucose not within range of 101 - 125 mg/dL
5. Use of prescription medications for diabetes or weight-loss
6. Use of and unwillingness to discontinue over the counter supplements (e.g. cinnamon, chromium, protein powders) or weight loss beverage or meal plans (e.g. SlimFast or Jenny Craig).
7. Low baseline albumin or pre-albumin levels (below normal reference range)
8. Significant anemia (Hemoglobin < 11 g/dL)
9. Known bleeding disorder or platelet dysfunction
10. Already eating a low protein diet (less than 14% total caloric intake from protein), as calculated from food diaries provided by subjects
11. Participating in intensive exercise training program (high to moderate intensity exercise greater than 210 minutes per week) or planning to start new exercise program during study period.
12. Significant co-morbidities (including kidney disease, liver disease, GI disease, cardiovascular disease, respiratory disease, malnutrition, substance abuse, psychiatric disease, or a diagnosed eating disorder).
13. Planned smoking cessation or attempt at smoking cessation during study period
14. Inability to tolerate meal replacement beverages due to palatability
15. Recent weight loss (> 5 lbs within 3 months).
16. Bariatric surgery, gastric banding or liposuction
17. Current or past (within 1 year) use of illicit drugs
18. Claustrophobia

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Reduction of BCAA intake | 3 months
  The principle outcome of this study is to determine if replacing 2/3rds of the subjects baseline protein intake with BCAA-free meal replacement beverages are a feasible method of selectively reducing BCAA consumption. Our principle outcome is to reduce BCAA intake by 50% or more in the Experimental Arm (BCAD2) of the study as compared to baseline intake.

SECONDARY OUTCOMES:
Weight | 3 months
  Weight in kg
Fat mass | 3 months
  Fat mass in kg
BMI | 3 months
  Weight in kg and height in meters will be combined to report BMI in kg/m^2
Resting metabolic rate | 3 months
  Resting metabolic rate in kcal/hour
Fasting blood glucose | 3 months
  Fasting blood glucose in mg/dL
Insulin | 3 months
  Insulin in ng/dL
HbA1c | 3 months
  HbA1c in mmol/mol
Glucose tolerance | 3 months
  Area under the curve in mg/dL/min

CONTACTS AND LOCATIONS:
Overall Officials: Dudley W Lamming, PhD, Principal Investigator — UW-Madison; Dawn B Davis, MD, PhD, Principal Investigator — UW-Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fontana L, Cummings NE, Arriola Apelo SI, Neuman JC, Kasza I, Schmidt BA, Cava E, Spelta F, Tosti V, Syed FA, Baar EL, Veronese N, Cottrell SE, Fenske RJ, Bertozzi B, Brar HK, Pietka T, Bullock AD, Figenshau RS, Andriole GL, Merrins MJ, Alexander CM, Kimple ME, Lamming DW. Decreased Consumption of Branched-Chain Amino Acids Improves Metabolic Health. Cell Rep. 2016 Jul 12;16(2):520-530. doi: 10.1016/j.celrep.2016.05.092. Epub 2016 Jun 23. PMID 27346343